CLINICAL TRIAL: NCT06555328
Title: Phase 2a Open-Label Basket Study to Evaluate Safety and Pharmacokinetics of INF904, an Oral C5aR1 Inhibitor, in Subjects With Moderate to Severe Chronic Spontaneous Urticaria or Hidradenitis Suppurativa
Brief Title: Evaluate Safety and Pharmacokinetics of INF904 in Subjects With Moderate to Severe Chronic Spontaneous Urticaria or Hidradenitis Suppurativa
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: InflaRx GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INF904- P2.1
Record Dates: First submitted 2024-08-07; First posted 2024-08-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Urticaria, Idiopathic; Hidradenitis; Hidradenitis Suppurativa
MeSH Terms: conditions — Chronic Urticaria; Hidradenitis; Hidradenitis Suppurativa | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1 CSU (Experimental): Lower dose of IFN904 BID
  Interventions: Drug: CSU lower dose treatment
- Arm 2 CSU (Experimental): Higher dose of IFN904 BID
  Interventions: Drug: CSU high dose treatment
- Arm 3 CSU (Experimental): Non responders IgE, higher dose of IFN904 BID
  Interventions: Drug: CSU non responders IgE - high dose treatment
- Arm 4 HS (Experimental): Lower dose of IFN904 BID
  Interventions: Drug: HS low dose treatment
- Arm 5 HD (Experimental): Medium dose of IFN904 BID
  Interventions: Drug: HS medium dose treatment
- Arm 6 HD (Experimental): High dose of IFN904 BID
  Interventions: Drug: HS high dose treatment

INTERVENTIONS:
Drug: CSU lower dose treatment — CSU lower dose treatment
  Arms: Arm 1 CSU
Drug: CSU high dose treatment — CSU high dose treatment
  Arms: Arm 2 CSU
Drug: CSU non responders IgE - high dose treatment — CSU non responders IgE - high dose treatment
  Arms: Arm 3 CSU
Drug: HS low dose treatment — HS low dose treatment
  Arms: Arm 4 HS
Drug: HS medium dose treatment — HS medium dose treatment
  Arms: Arm 5 HD
Drug: HS high dose treatment — HS high dose treatment
  Arms: Arm 6 HD

SUMMARY:
The study duration for an individual subject includes screening (14 days), the treatment period (28 days) and the observational follow-up period of 28 days, in total 70 days ± 6 days. All subjects will receive IMP for 28 days followed by one End of Study (EOS) visit, 4 weeks after EOT visit.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Subjects must be 18 years or older at the time of signing the informed consent.

Exclusion Criteria:

* Subjects with known severe or life-threatening hypersensitivity reaction to any other CSU/HS treatment according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE).
* Subjects who have any other skin disease that may interfere with assessment of CSU or HS.
* Subjects who have an active infection or history of infection(s) as follows:

  1. Any infection requiring systemic treatment within 14 days prior to baseline.
  2. A history of opportunistic, recurrent, or chronic infections that, in the opinion of the Investigator, might cause this study to be detrimental to the subject.
* Subjects with known progressed liver disease (Child-Pugh B or C)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-01-22 (Actual); Study Completion 2026-01-22 (Actual)

PRIMARY OUTCOMES:
Frequency, severity, and relatedness of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs). | Through study completion, an average of 10 weeks
  Frequency, severity, and relatedness of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) using MedDRA classification.

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | Through study completion, an average of 10 weeks
  Plasma PK parameters of INF904
Minimum Plasma Concentration [Cmin] | Through study completion, an average of 10 weeks
  Plasma PK parameters of INF904
Time of occurrence of maximum plasma concentration [tmax] | Through study completion, an average of 10 weeks
  Plasma PK parameters of INF904
Systemic exposure, defined as the Area Under the Curve [AUC0-24] | Through study completion, an average of 10 weeks
  Plasma PK parameters of INF904
Systemic exposure, defined as the Area Under the Curve [AUClast] | Through study completion, an average of 10 weeks
  Plasma PK parameters of INF904

CONTACTS AND LOCATIONS:
Locations (29):
- United States (9):
  - First OC Dermatology Research Inc., Fountain Valley, California
  - Ziaderm Research LLC, North Miami Beach, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Kentucky Advanced Medical Research LLC, Murray, Kentucky
  - MediSearch LLC, Saint Joseph, Missouri
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Wright State Physicians, Fairborn, Ohio
  - Progressive Clinical Research, PA, Texas City, Texas
- Bulgaria (5):
  - Medical Center Medconsult, Pleven OOD, Lovech
  - Medical Center Medconsult pleven OOD, Pleven
  - Medical Center Etika, Plovdiv
  - ASMC IPSMC Skin and Venereal Diseases,, Sofia
  - Medical Center Excelsior OOD,, Sofia
- Georgia (4):
  - LTD "Health", Batumi
  - LTD "Israel-Georgian Medical Research Clinic Healthycore", Tbilisi
  - LLC "Center of Allergy and Immunology", Tbilisi
  - LLC "Aversi Clinic", Tbilisi
- Germany (5):
  - "Institut Allergieforschung Charité - Universitatsmedizin Berlin", Berlin
  - Katholisches Klinikum Bochum gGmbH/ St.Josef-Hospital Bochum, Dermatologie, Bochum
  - Universitatsklinikum Dresden Carl Gustav Carus, Dresden
  - Universitätsklinikum Frankfurt, Klinik für Dermatologie, Venerologie und Allergologie, Frankfurt
  - "Klinikum der Universitat (LMU) Klinik und Poliklinik far Dermatologie und Allergologie", München
- Greece (2):
  - General University Hospital "Attikon", Athens
  - General Hospital of Thessaloniki "Papageorgiou", Thessaloniki
- Poland (4):
  - Klinika Dermatologii, Wenerologii i Alergologii, UNIWERSYTECKIE CENTRUM KLINICZNE, ul., Gdansk
  - Oddziat Kliniczny Wewnetrznych, Astmy i Alergii z Odcinkiem dla Dzieci, Samodzielny Publiczny Zaktad Opieki Zdrowotnej Uniwersytecki Szpital Kliniczny, Lodz
  - Labderm Essence sp., Ossy
  - "Cityclinic Przychodnia Lekarsko-Psychologiczna Matusiak Spolka Partnerska", Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided